CLINICAL TRIAL: NCT05439629
Title: A Multicenter, Randomized, Double-blind Phase III Clinical Study Comparing the Efficacy and Safety of BAT5906 and Ranibizumab (Lucentis®) in Patients With Neovascular Age-related Macular Degeneration
Brief Title: Efficacy Evaluation Study of BAT5906 and Lucentis® in Patients With Macular Degeneration
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bio-Thera Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BAT5906-004-CR
Record Dates: First submitted 2022-06-13; First posted 2022-06-30 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Neovascular (Wet) Age-related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group：BAT5906 (Experimental): Intravitreal injection; Dosage: 4.0 mg / eye / time, 50 μl; Duration of administration: every 4 weeks, administered to week 48, not administered at 52 weeks.
  Interventions: Drug: BAT5906 injection
- Control group：Lucentis® (Active Comparator): Intravitreal injection; Dosage: 0.5 mg / eye / time, 50 μl; Duration of administration: every 4 weeks, administered to week 48, not administered at 52 weeks.
  Interventions: Drug: Lucentis

INTERVENTIONS:
Drug: BAT5906 injection — 4.0 mg/eye/time, 50 μl, intravitreal injection
  Arms: Experimental group：BAT5906
Drug: Lucentis — 0.5 mg/eye/time, 50 μl, intravitreal injection
  Arms: Control group：Lucentis®

SUMMARY:
A non-inferiority design was used to conduct a randomized, double-blind, parallel-controlled multi-center study. A total of 488 subjects with neovascular (wet) age-related macular degeneration (w-AMD) were planned to be enrolled. Qualified subjects were divided into experimental group and control group in a 1:1 ratio, and stratified randomized according to the letter value of baseline period and whether the eyes had received anti-VEGF drug treatment. The experimental group received BAT5906 injection. The control group received Lucentis® treatment. Only 1 eye per subject was included in this study.

DETAILED DESCRIPTION:
A non-inferiority design was used to conduct a randomized, double-blind, parallel-controlled multi-center study. A total of 488 subjects with neovascular (wet) age-related macular degeneration (w-AMD) were planned to be enrolled. Qualified subjects were divided into experimental group and control group in a 1:1 ratio, and stratified randomized according to the letter value of baseline period and whether the eyes had received anti-VEGF drug treatment. The experimental group received BAT5906 injection. The control group received Lucentis® treatment. Only 1 eye per subject was included in this study.

The administration regimen was as follows: once every 4 weeks, 4mg BAT5906 or 0.5mg Lucentis® were injected intravitreal each time, the treatment period of the study was 48 weeks, a total of 13 administration times, the last follow-up was conducted at the 52nd week, the last visit did not require treatment, only efficacy and safety assessment, and blood samples were collected as required.

Ophthalmic examination, vital signs, physical examination, and laboratory examination were performed for efficacy and safety assessment according to the test procedures specified in the protocol, and blood samples were collected for immunogenicity indicators. Change in best corrected visual acuity (BCVA) from baseline was assessed by ETDRS visual acuity chart at 4-week intervals. The primary efficacy measure was the change in BCVA from baseline at 52 weeks. Secondary efficacy measures were the change in best corrected visual acuity (BCVA) of the target eye from baseline and the change in macular fovea thickness (CRT) from baseline at weeks 12, 24, 36 and 48.

Blood samples were collected according to the time points specified in the program, and the serum anti-drug antibody (ADA) was detected. Titer analysis and neutralizing antibody (Nab) analysis were performed on the samples confirmed as positive by ADA.

A non-inferiority design was used to conduct a randomized, double-blind, parallel-controlled multi-center study. A total of 488 subjects with neovascular (wet) age-related macular degeneration (w-AMD) were planned to be enrolled. Qualified subjects were divided into experimental group and control group in a 1:1 ratio, and stratified randomized according to the letter value of baseline period and whether the eyes had received anti-VEGF drug treatment. The experimental group received BAT5906 injection. The control group received Lucentis® treatment. Only 1 eye per subject was included in this study.

The administration regimen was as follows: once every 4 weeks, 4mg BAT5906 or 0.5mg Lucentis® were injected intravitreal each time, the treatment period of the study was 48 weeks, a total of 13 administration times, the last follow-up was conducted at the 52nd week, the last visit did not require treatment, only efficacy and safety assessment, and blood samples were collected as required.

Ophthalmic examination, vital signs, physical examination, and laboratory examination were performed for efficacy and safety assessment according to the test procedures specified in the protocol, and blood samples were collected for immunogenicity indicators. Change in best corrected visual acuity (BCVA) from baseline was assessed by ETDRS visual acuity chart at 4-week intervals. The primary efficacy measure was the change in BCVA from baseline at 52 weeks. Secondary efficacy measures were the change in best corrected visual acuity (BCVA) of the target eye from baseline and the change in macular fovea thickness (CRT) from baseline at weeks 12, 24, 36 and 48.

Blood samples were collected according to the time points specified in the program, and the serum anti-drug antibody (ADA) was detected. Titer analysis and neutralizing antibody (Nab) analysis were performed on the samples confirmed as positive by ADA.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and sign the informed consent, and be willing to follow up according to the time specified in the trial;
2. Age 50-85 years old (including boundary value), male and female;
3. Study the subjects who were diagnosed with neovascular age-related macular degeneration and still had active lesions confirmed by imaging examination. Active lesions were defined as the presence of any of the following lesions in the macular area: ① intraretinal fluid; ② Lipid exudation in the retina; ③ Subretinal fluid; (4) Subretinal hemorrhage; (5) Retinal pigment epithelium detachment; ⑥ Choroidal neovascularization leakage;
4. The total area of the study eye lesions ≤30mm2(12 optic disc areas) was confirmed by the film reading center before randomization;
5. The BCVA of the study eye at screening and baseline was 73-19 letters (ETDRS visual acuity chart, including boundary values), equivalent to Snellen visual acuity 20/40 to 20/400;
6. BCVA≥19 letters, equivalent to Snellen visual acuity ≥20/400, measured by ETDRS visual chart at screening and baseline in non-study eyes.

Exclusion Criteria:

1. The study eyes received any intravitreal anti-VEGF therapy (such as bevacizumab, abbercept, ranibizumab, conbercept, etc.) within 3 months before randomization;
2. The study eyes had received the following treatments within 3 months before randomization: verteporfin photodynamic therapy (PDT), macular laser photocoagulation, transpillary thermotherapy (TTT), and other surgeries for AMD;
3. The study eyes had undergone the following ophthalmic surgeries: vitrectomy, anti-glaucoma surgery, and macular transposition. The study eyes had undergone internal eye surgery (including cataract surgery) within 3 months before randomization, or external eye surgery within 1 month before randomization;
4. The study eyes received intravitreal injection treatment (such as triamcinolone acetonide and dexamethasone) within 3 months before randomization, intravitreal injection of dexamethasone sustained release within 6 months, and injection of long-acting corticosteroids (such as triamcinolone acetonide, etc.) within, periocular or subconjunctival injection of any eye 3 months before randomization;
5. Study eyes with ocular diseases affecting central vision (such as diabetic retinopathy, retinal vein occlusion, uveitis, vascular striation, pathological myopia, retinal detachment, macular hole, macular epiretinal membrane, toxoplasmosis, optic nerve diseases);
6. Study eyes with foveal ground pattern atrophy, scar or fibrosis, dense subfoveal hard exudation, retinal pigment epithelium (RPE) tear involving the center of the macula (confirmed by the reading center during screening);
7. The study eyes had choroidal neovascularization not caused by nAMD, progressive retinopathy affecting corrected visual acuity, and any eye had vitreous hemorrhage or a history of vitreous hemorrhage, or a history of retinal detachment;
8. The equivalent spherical mirror of the study eye with refractive error showed more than -6.0 diopters. For patients with previous refractive surgery or cataract surgery, the preoperative refractive error of the study eye should not exceed -6.0 diopters;
9. The study eyes were lens free (excluding IOL eyes) or posterior lens capsule rupture (except YAG laser posterior capsuleotomy after IOL implantation more than 1 month before screening);
10. The study eye has obvious refractive interstitial opacity or pupil failure, including cataract and corneal opacity, which may interfere with visual acuity assessment, safety assessment or fundus photography;
11. The study eyes had pupil afferent defect (APD);
12. Study eyes had uncontrolled glaucoma at randomization, defined as intraocular pressure that remained higher than 25mmHg after medical treatment or as judged by the investigator;
13. Non-study eyes received photodynamic therapy (PDT) within 1 month before randomization;
14. History of idiopathic or autoimmune associated uveitis in any eye;
15. Pseudocyst stripping syndrome in any eye;
16. Active eye infection in any eye (e.g., blepharitis, infectious conjunctivitis, keratitis, scleritis, iridecocyclitis, endophthalmitis);
17. Systemic drugs that cause crystal or retinal toxicity, such as deferoxamine, chloroquine/hydroxychloroquine, phenothiazine and ethambutol or tamoxifen, are currently being used or may be required;
18. Allergic reaction or history to sodium fluorescein and indocyanine green, allergic history to protein products for therapeutic or diagnostic use, or known allergic reaction to any monoclonal antibody;
19. Patients who had surgery within 1 month before randomization and the surgery did not heal, and the investigator judged that the study drug had an effect on healing;
20. Presence of clinically significant active systemic infectious disease under treatment;
21. History of myocardial infarction, unstable angina, coronary revascularization, cerebrovascular accident (including TIA), other thromboembolic diseases (such as thromboembolic angiitis, pulmonary embolism, deep vein thrombosis, portal vein thrombosis, etc.), New York Heart Association (NYHA) grade ≥II cardiac dysfunction within 6 months before randomization, Severe unstable ventricular arrhythmias;
22. Patients with active disseminated intravascular coagulation and significant bleeding tendency (such as hemoptysis, hematemesis, severe purpura, etc.) within 3 months before randomization, or who had received anticoagulant and antiplatelet therapy other than aspirin /NSAIDs within 14 days before screening;
23. Poorly controlled hypertension before randomization (defined as sitting systolic blood pressure ≥160mmHg or diastolic blood pressure ≥100mmHg after antihypertensive medication);
24. Any uncontrollable clinical problems (such as serious mental, neurological, cardiovascular, respiratory and other system diseases and malignant tumors);
25. Abnormal liver and kidney function (ALT and AST should not be higher than 2.5 times of the upper limit of normal value in the central laboratory; Crea and BUN shall not be higher than 2 times of the upper limit of normal value in the central laboratory);
26. Abnormal coagulation function (prothrombin time > upper limit of normal 3 seconds or activated partial thromboplastin time > upper limit of normal 10 seconds);
27. Patients with any of the following infections: active hepatitis B (HBV DNA > 1000 IU/mL if HBsAg(+)), hepatitis C, AIDS, or syphilis (syphilis RPR confirmatory test positive);
28. Planned parenthood during pregnancy or lactation, or during the study period and within 6 months after the study. The pregnancy test of fertile female patients was positive during the screening period;
29. Subjects who have participated in any drug (excluding vitamins and minerals) in the clinical trial within 3 months before randomization and have been treated with the experimental drug or device;
30. The researcher believes that it is not suitable for this study.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 488 (Actual)
Dates: Start 2022-07-07 (Actual); Primary Completion 2025-04-22 (Actual); Study Completion 2025-04-22 (Actual)

PRIMARY OUTCOMES:
The change in the BCVA value | Week 52
  Compared to baseline, two groups of subjects studied the value of changes in ocular 52nd week BCVA
The change in the BCVA value | at weeks 12, 24, 36, and 48
  Compared to baseline, two groups of subjects studied the changes in bcVA at weeks 12, 24, 36, and 48 of the eye
BCVA increased the proportion of subjects with >10, >15, ≥30 words | in the 24th and 52nd weeks
  Compared with baseline, the proportion of subjects with 30 words of BCVA in the 24th and 52nd weeks of the study eye was improved > 10, >15, ≥ 30 words;
BCVA reduced the proportion of subjects < 10, < 15 words | at weeks 24 and 52
  Compared with baseline, the proportion of subjects in both groups who studied eye bcVA at weeks 24 and 52 decreased <10, < 15 words
Changes in the thickness of the macular fovea (CRT). | at weeks 12, 24, 36, 48, and 52
  Changes in the thickness of the macular fovea (CRT) at weeks 12, 24, 36, 48, and 52 were studied in both groups of subjects compared to baseline

SECONDARY OUTCOMES:
Vital signs | Weeks 1 to 52
  Number of participants with abnormal vital signs
physical examination | Weeks 1 to 52
  Number of participants with abnormal physical examination findings
Laboratory tests | Weeks 1 to 52
  Number of participants with abnormal laboratory test results
electrocardiogram（ ECG ） | Weeks 1 to 52
  Number of participants with abnormal ECG readings
Antibiotic antibodies (ADA) | Weeks 1 to 52
  Resistance antibody (ADA) situation in the subject
Adverse events（AE） | Weeks 1 to 52
  Ocular and non-ocular adverse events (AE) and serious adverse events (SAE)
Adverse events of particular concern (possible adverse reactions to the eye) | Weeks 1 to 52
  Endophthalmia, increased intraocular pressure, subconjunctival hemorrhage, ocular foreign body sensation, visual impairment, corneal abrasions, lens damage, retinal detachment, retinal artery occlusion, etc.; Possible systemic adverse effects include non-ocular bleeding, increased blood pressure, and thromboembolic events

OTHER OUTCOMES:
Immunogenicity evaluation | Weeks 1 to 52
  Blood samples from BAT5906 and Lucentis® injections were detected for ADA detection and analysis to detect anti-BAT5906 antibodies (ADA). Serum antibodies (ADA) are tested, and neutralizing antibody (Nab) analysis will continue if the ADA is confirmed positive.

CONTACTS AND LOCATIONS:
Overall Officials: Youxin Chen, Doctor, Principal Investigator — Peking Union Medical College; Xiaolin Liu, Doctor, Principal Investigator — Affiliated Optometry Hospital of Wenzhou Medical University; Mingwei Zhao, Doctor, Principal Investigator — Peking University People's Hospital; Yi Chen, Doctor, Principal Investigator — China-Japan Friendship Hospital; Hong Dai, Doctor, Principal Investigator — Beijing Hospital; Yong Tao, Doctor, Principal Investigator — Beijing Chao Yang Hospital; Linna Lu, Doctor, Principal Investigator — The Ninth People's Hospital Affiliated to Shanghai Jiao Tong University School of Medicine; Hongping Cui, Doctor, Principal Investigator — Shanghai Oriental Hospital; Xiaolin Liang, Doctor, Principal Investigator — Sun Yat-sen Ophthalmic Center, Sun Yat-sen University; Pengxia Wan, Doctor, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University; Yuqing Lan, Doctor, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University; Haoyu Chen, Doctor, Principal Investigator — Shantou University-Chinese University of Hong Kong Joint Shantou International Eye Centre; Xiyuan Zhou, Doctor, Principal Investigator — The Second Affiliated Hospital of Chongqing Medical University; Xiaohong Meng, Doctor, Principal Investigator — The First Affiliated Hospital of Army Medical University (Southwest Hospital); Jinglin Yi, Doctor, Principal Investigator — The Affiliated Eye Hospital of Nanchang University; Hongmei Zheng, Doctor, Principal Investigator — People's Hospital of Wuhan University (Hubei Provincial People's Hospital); Liuhua Tong, Doctor, Principal Investigator — People's Hospital of Quzhou; Zongming Song, Doctor, Principal Investigator — Henan Eye Center (Henan Eye Hospital); Shenzhi Liang, Doctor, Principal Investigator — The First Affiliated Hospital of Zhengzhou University; Junfeng Mao, Doctor, Principal Investigator — Xiangya Hospital of Central South University; Xiangwen Shu, Master, Principal Investigator — Jinan Second People's Hospital; Yuanbin Li, Doctor, Principal Investigator — Yantai Yuhuangding Hospital; Shanjun Cai, Doctor, Principal Investigator — Zunyi Medical College; Xian Wang, Doctor, Principal Investigator — Affiliated Hospital of Guizhou Medical University; Xu Li, Master, Principal Investigator — The Fourth People's Hospital of Shenyang; Rongrong Zhu, Bachelor, Principal Investigator — Affiliated Hospital of Nantong University; Wei Wei, Doctor, Principal Investigator — Jiangsu Provincial Hospital of Traditional Chinese Medicine; Yabin Sun, Doctor, Principal Investigator — The First Hospital of Jilin University; Liming Tao, Doctor, Principal Investigator — The Second Hospital of Anhui Medical University; Hongjian Ma, Doctor, Principal Investigator — Aier Eye Hospital, Guangzhou; Yaohong Wu, Doctor, Principal Investigator — Second Hospital of Shanxi Medical University; Jian Guo, Doctor, Principal Investigator — First Affiliated Hospital of Fujian Medical University; Xiaoling Luo, Doctor, Principal Investigator — Shenzhen People's Hospital; Qiuhong Liu, Doctor, Principal Investigator — The First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine; Xinquan Liu, Doctor, Principal Investigator — Shanghai University of Traditional Chinese Medicine; Lifei Wang, Doctor, Principal Investigator — Hebei Provincial Eye Hospital; Dan Zhu, Doctor, Principal Investigator — The Affiliated Hospital of Inner Mongolia Medical University; Xuemei Pan, Master, Principal Investigator — The Affiliated Eye Hospital of Shandong University of Chinese Medicine; Yanfei Qiu, Doctor, Principal Investigator — Pingxiang People's Hospital; Zhen Zhang, Doctor, Principal Investigator — Xuzhou Central Hospital; Jingbo Li, Doctor, Principal Investigator — Luoyang Third People's Hospital; Xinyan Xu, Master, Principal Investigator — Weifang Eye Hospital; Lan Li, Master, Principal Investigator — The First People's Hospital of Kunming; Hongxia Yang, Bachelor, Principal Investigator — Jinzhong First People's Hospital; Miaoqin Wu, Doctor, Principal Investigator — Zhejiang Provincial People's Hospital; Zhaozeng Lu, Doctor, Principal Investigator — Huashan Hospital; Gangfeng Cui, Doctor, Principal Investigator — Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University; Quanyong Yi, Doctor, Principal Investigator — Ningbo Eye Hospital; Ruifeng Wang, Doctor, Principal Investigator — The Second People's Hospital of Zhengzhou
Locations (48):
- China (48):
  - Affiliated Hospital of Inner Mongolia Medical University, Beijing
  - Beijing Chao Yang Hospital, Beijing
  - Beijing Hospital, Beijing
  - China-Japan Friendship Hospital, Beijing
  - Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing
  - Peking University People's Hospital, Beijing
  - Xiangya Hospital of Central South University, Changsha
  - The First Affiliated Hospital of Army Medical University (Southwest Hospital), Chongqing
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing
  - First Affiliated Hospital of Fujian Medical University, Fujian
  - First Affiliated Hospital, Sun Yat-Sen University, Guangzhou
  - Guangzhou Aier Eye Hospital, Guangzhou
  - Sun Yat-sen Ophthalmic Center, Sun Yat-sen University, Guangzhou
  - The First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine, Guangzhou
  - Affiliated Hospital of Guizhou Medical University, Guiyang
  - Zhejiang Provincial People's Hospital, Hangzhou
  - The Second Hospital of Anhui Medical University, Hefei
  - People's Hospital of Wuhan University (Hubei Provincial People's Hospital), Hubei
  - The First Hospital of Jilin University, Jilin
  - Jinan Second People's Hospital, Jinan
  - The Affiliated Eye Hospital of Shandong University of Chinese Medicine, Jinan
  - Jinzhong First People's Hospital, Jinzhong
  - The First People's Hospital of Kunming, Kunming
  - Luoyang Third People's Hospital, Luoyang
  - The Affiliated Eye Hospital of Nanchang University, Nanchang
  - Jiangsu Provincial Hospital of Traditional Chinese Medicine, Nanjing
  - Affiliated Hospital of Nantong University, Nantong
  - Ningbo Eye Hospital, Ningbo
  - Pingxiang People's Hospital, Pingxiang
  - People's Hospital of Quzhou, Quzhou
  - Huashan Hospital, Shanghai
  - Shanghai Oriental Hospital, Shanghai
  - Shanghai University of Traditional Chinese Medicine, Shanghai
  - The Ninth People's Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai
  - Shantou University-Chinese University of Hong Kong Joint Shantou International Eye Centre, Shantou
  - The Fourth People's Hospital of Shenyang, Shenyang
  - Shenzhen People's Hospital, Shenzhen
  - Second Hospital of Shanxi Medical University, Taiyuan
  - Taizhou Hospital of Zhejiang Province, Taizhou
  - Weifang Eye Hospital, Weifang
  - Wenzhou Medical University Affiliated Optometry Hospital, Wenzhou
  - Hebei Provincial Eye Hospital, Xingtai
  - Xuzhou Central Hospital, Xuzhou
  - Yantai Yuhuangding Hospital, Yantai
  - Henan Eye Center (Henan Eye Hospital), Zhengzhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou
  - The Second People's Hospital of Zhengzhou, Zhengzhou
  - Zunyi Medical College, Zunyi

IPD SHARING:
Plan to Share IPD: No